CLINICAL TRIAL: NCT00533936
Title: Adjuvant Trastuzumab vs Observation in Locally Advanced Breast Cancer Treated With Neoadjuvant Trastuzumab
Brief Title: Trastuzumab or Observation After Combination Chemotherapy and Trastuzumab in Treating Patients Undergoing Surgery for Stage II or Stage III Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000557417; MEX-INC-INCAN-CC-09506
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide; Doxorubicin; Fluorouracil; Paclitaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: trastuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: paclitaxel
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with trastuzumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving trastuzumab after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether trastuzumab is more effective than observation when given after combination chemotherapy and trastuzumab in treating patients with breast cancer.

PURPOSE: This randomized phase II trial is studying trastuzumab to see how well it works compared with observation when given after combination chemotherapy and trastuzumab in treating patients undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the percentage of pathological responses in patients with stage II or III breast cancer treated with neoadjuvant therapy comprising fluorouracil, doxorubicin hydrochloride, and cyclophosphamide followed by trastuzumab (Herceptin®) and paclitaxel.
* To compare the disease-free survival of patients treated with adjuvant therapy comprising trastuzumab versus observation.

Secondary

* To measure the overall survival at 3 years in these patients.
* To measure the cardiac safety profile of these regimens in these patients.
* To measure the percentage of patients that become negative on the fluorescence in situ hybridization (FISH) test at the end of neoadjuvant therapy.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I :

  * Neoadjuvant therapy: Patients receive fluorouracil IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab (Herceptin®) IV over 30-90 minutes and paclitaxel IV over 1 hour once a week for 12 weeks.

After completion of neoadjuvant therapy, patients proceed to surgery.

* Surgery: Patients undergo definitive surgery. Some patients may also undergo radiotherapy*.

NOTE: *Patients with initial tumor > 5 cm, inflammatory breast cancer, or with a skin condition or final pathological evaluation of metastasis to > 4 nodes or 1-3 nodes with capsular ruptures or extension to fatty tissues receive adjuvant radiotherapy.

* Adjuvant therapy: Beginning 4 weeks after surgery, patients receive trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for 13 courses.

  * Arm II:
* Neoadjuvant therapy: Patients receive neoadjuvant therapy as in arm I.
* Surgery: Patients undergo definitive surgery. Some patients may also undergo radiotherapy if clinically indicated.
* Observation: Beginning 4 weeks after surgery, patients undergo observation. In both arms, patients with estrogen receptor- and/or progesterone receptor-positive disease also receive anastrozole daily for 5 years. Premenopausal patients with remaining ovarian function (as confirmed by follicle-stimulating hormone [FSH] and estradiol) after completion of anastrozole undergo chemical or surgical ovarian ablation.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then once a year thereafter.

PROJECTED ACCRUAL: A total of 160 patients (80 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer by needle biopsy

  * Diagnosed within the past 4 weeks
  * Clinical stage IIB, IIIA, IIIB, or IIIC disease
* Palpable adenopathies present
* HER2/neu-positive disease, as evidenced by either of the following:

  * HER2/neu overexpression (3+) by immunohistochemistry (IHC)
  * HER2/neu amplification by fluorescence in situ hybridization (FISH)
* No metastatic disease by chest radiography, hepatic ultrasound, and bone scan (metastatic bone series if no nuclear medicine is available)
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor status known

PATIENT CHARACTERISTICS:

* Premenopausal or postmenopausal
* WHO performance status 0-2
* Not pregnant or nursing
* Normal hepatic, renal, and hematological function
* LVEF ≥ 55% by nuclear medicine study or echocardiogram
* No prior history of cancer, except carcinoma in situ of the cervix
* No allergic reaction or hypersensitivity to paclitaxel and/or trastuzumab (Herceptin®)

PRIOR CONCURRENT THERAPY:

* No prior cancer therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of pathological responses
Disease-free survival

SECONDARY OUTCOMES:
Overall survival at 3 years
Cardiac toxicity
Percentage of patients that become negative on the fluorescence in situ hybridization (FISH) test at the end of neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Arce-Salinas, MD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital General de Mexico, Mexico City, Mexico City